CLINICAL TRIAL: NCT02145247
Title: Ovarian Morphology and Theca Cell Androgen Production in Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Professor, Reproductive Endocrinology. Fellowship Director, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UCSD-140260
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal adult women (Active Comparator): 1. Images of the both ovaries will be obtained using vaginal ultrasound and the number, size, and spatial arrangement of ovarian follicles will be noted for both ovaries in each subject.
  2. On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  3. Blood samples will be obtained at T = -0.5, 0, and +24 hours.
  4. Blood sample will be used for DNA testing to identify genes that may be associated with androgen production.
  5. One to two weeks after hCG stimulation testing each subject will come to the CTRI for an Oral Glucose Tolerance Test (OGTT). Each subject will ingest 75 gm of a glucose solution and blood samples will be obtained at 0, 15, 30, 60, 120 and 180 minutes after the glucose load.
  Interventions: Drug: hCG
- Women with PCOS (Active Comparator): 1. Images of the both ovaries will be obtained using vaginal ultrasound and the number, size, and spatial arrangement of ovarian follicles will be noted for both ovaries in each subject.
  2. On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  3. Blood samples will be obtained at T = -0.5, 0, and +24 hours.
  4. Blood sample will be used for DNA testing to identify genes that may be associated with androgen production.
  5. One to two weeks after hCG stimulation testing each subject will come to the CTRI for an Oral Glucose Tolerance Test (OGTT). Each subject will ingest 75 gm of a glucose solution and blood samples will be obtained at 0, 15, 30, 60, 120 and 180 minutes after the glucose load.
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG — 3. On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  4. Blood samples will be obtained at T = -0.5, 0, and +24 hours.
  Other Names: Re-combinant human choriogonadotropin

SUMMARY:
Women with PCOS suffer from excess male hormone (androgen) production by the ovary. Androgen is made by cells that surround follicles that contain eggs. As the follicles (and eggs) grow and mature, there are more androgen producing cells. Women with PCOS have more follicles than normal women and therefore more androgen producing cells. While androgen production has been associated with the number of follicles, the relationship to the individual size of follicles in PCOS or normal women. This study intends to determine whether the size and number of ovarian follicles are correlated to androgen production in PCOS and normal women.

DETAILED DESCRIPTION:
In women with polycystic ovary syndrome (PCOS), the major abnormality is excessive ovarian androgen production marked by increased serum testosterone (T) and androstenedione (A) levels. Studies to determine the alteration in ovarian steroidogenesis that lead to abnormal production of ovarian androgens have revealed increased CYP17 gene expression with accentuated 17-hydroxylase activity leading to exaggerated 17-hydroxyprogesterone (17P) responses to LH stimulation. In contrast, T and A responses did not distinguish between PCOS and normal women, although these androgens were clearly greater in the former compared to the latter group. As a result, 17P responsiveness has been employed to determine the functional capacity of the ovary to produce androgen. Stimulatory agents have included GnRH agonist, Lupron, at a dose of 10 microgram per kilogram, or hCG at a dose of 10,000 IU.

The investigators recently showed that hCG administered intravenously in a dose-response fashion revealed gradual increases of 17P and a non-dose dependent increase of serum T and A. The pattern of steroid hormone production revealed the predominant pathway by which androgens are generated in women with PCOS. Extending these studies, the investigators selected the mid-maximal dose of hCG to stimulate ovarian androgens and included morphometric measures of the ovary, such as ovarian follicle number (as determined by ultrasound) and related hormones, such as anti-mullerian hormone and inhibin B, both products of the ovarian follicle. The results showed that increased androgen and 17P responses in PCOS women were associated with increased antral follicle number and greater AMH levels compared to normal women. Inhibin B levels were similar between groups.

Based on responses observed in normal women, the PCOS women were divided into two groups. Those with 17P responses that did not exceed the normal mean plus 2 standard deviations (normal responder PCOS; NR-PCOS) and those that did exceed the normal response (high responder PCOS; HR-PCOS). This separation occurred at a rate of 50%. Notably, serum AMH levels were 2-fold higher in NR-PCOS compared to HR-PCOS. This finding was puzzling as serum AMH levels have been shown to correlate to the number of small follicles present in ovaries suggesting that AMH may be a surrogate for small follicle number. However, both PCOS subgroups had equivalent follicle numbers. The investigators hypothesize that the NR-PCOS have greater number of small follicles compared to HR-PCOS. To address this issue the investigators propose to assess the number of small follicles in NR- and HR-PCOS women and normal controls.

In a secondary consideration the HR-PCOS group was heavier than the NR-PCOS. This implies that the HR-PCOS women may have had greater insulin resistance and hyperinsulinemia that may have contributed to the significantly higher 17P responses to hCG. As a result, the investigators will also perform an oral glucose tolerance test in all subjects.

Power Analysis Results of the investigators' pilot study have shown that approximately 50% of PCOS women will exhibit 17OHP responses to hCG stimulation similar to those of normal women. Consequently, a sample size of 20 subjects in each group has an 80% power to detect a difference in the means of 0.820 ng/ml (the difference between the average 17OHP expression level in high responder PCOS women (HR-PCOS), 2.840 ng/ml, and that of normal responder PCOS (NR-PCOS) women, 2.02 ng/ml), which is a 33% increase. In the proposed study, the investigators believe that HR-PCOS (n=20) will show significantly greater (33% more) 17OHP production in response to hCG stimulation than NR-PCOS (n=20) at a power of 0.8 and a type I error rate of 0.05. The investigators will recruit 25 subjects in each group to allow for subject drop out. A secondary analysis will be performed between women with PCOS and normal controls (n=20).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be determined to have PCOS based on clinical history of irregular menses and clinical or laboratory evidence of hyperandrogenism and polycystic ovaries on ultrasound
2. Subjects should not have been on any hormonal therapy or metformin for at least 2 months prior to study start
3. Subjects will be determined to be normal controls if they have a clinical history of regular periods

Exclusion Criteria:

1. Women with hemoglobin less than 11 gm/dl at screening evaluation
2. Women with untreated thyroid abnormalities
3. Pregnant women or women who are nursing
4. Women with BMI > 37
5. Women with known sensitivity to the agents being used
6. Women with diabetes, or renal, liver, or heart disease

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Jeffrey Chang, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Rosencrantz MA, Coffler MS, Haggan A, Duke KB, Donohue MC, Shayya RF, Su HI, Chang RJ. Clinical evidence for predominance of delta-5 steroid production in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Apr;96(4):1106-13. doi: 10.1210/jc.2010-2200. Epub 2011 Jan 26. PMID 21270326
- [Background] Pigny P, Jonard S, Robert Y, Dewailly D. Serum anti-Mullerian hormone as a surrogate for antral follicle count for definition of the polycystic ovary syndrome. J Clin Endocrinol Metab. 2006 Mar;91(3):941-5. doi: 10.1210/jc.2005-2076. Epub 2005 Dec 20. PMID 16368745
- [Background] Dewailly D, Gronier H, Poncelet E, Robin G, Leroy M, Pigny P, Duhamel A, Catteau-Jonard S. Diagnosis of polycystic ovary syndrome (PCOS): revisiting the threshold values of follicle count on ultrasound and of the serum AMH level for the definition of polycystic ovaries. Hum Reprod. 2011 Nov;26(11):3123-9. doi: 10.1093/humrep/der297. Epub 2011 Sep 16. PMID 21926054
- [Background] Laven JS, Mulders AG, Visser JA, Themmen AP, De Jong FH, Fauser BC. Anti-Mullerian hormone serum concentrations in normoovulatory and anovulatory women of reproductive age. J Clin Endocrinol Metab. 2004 Jan;89(1):318-23. doi: 10.1210/jc.2003-030932. PMID 14715867

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Adult Women; Women With PCOS: 1. Images of the both ovaries will be obtained using vaginal ultrasound and the number, size, and spatial arrangement of ovarian follicles will be noted for both ovaries in each subject.
  2. On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  3. Blood samples will be obtained at T = -0.5, 0, and +24 hours.
  4. Blood sample will be used for DNA testing to identify genes that may be associated with androgen production.
  5. One to two weeks after hCG stimulation testing each subject will come to the CTRI for an Oral Glucose Tolerance Test (OGTT). Each subject will ingest 75 gm of a glucose solution and blood samples will be obtained at 0, 15, 30, 60, 120 and 180 minutes after the glucose load.
  hCG: 3. On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  4. Blood samples will be obtained at T = -0.5, 0, and +24 hours.
Period: Overall Study
Arm/Group | Normal Adult Women | Women With PCOS
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Adult Women | Women With PCOS | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Full Range); unit: years] | 26.9 [19 to 34] | 26.3 [19 to 37] | 26.6 [19 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39
Sex and gender [Count of Participants; unit: Participants] | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of 17-OHP Levels From Baseline
Description: On study day one, recombinant-hCG (r-hCG) will be administered intravenously at a dose of 25 micrograms.
  Blood samples will be obtained before and after r-hCG adminstration
Time Frame: before and 24 hours after adminisration of r-hCG
Population: Normal adult women and adult women with PCOS
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Normal Adult Women | Women With PCOS
Number analyzed (Participants) | 20 | 19
percent change | 67 (10) | 140 (26)

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no untoward or unfavorable medical occurrences in participating subjects.
Arm/Group | Normal Adult Women | Women With PCOS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT02145247/Prot_SAP_000.pdf